CLINICAL TRIAL: NCT02807064
Title: Evaluation of the Effectiveness of Treatment With Bifidobacteria in Children Affected by Seasonal Allergic Rhinitis
Brief Title: Effectiveness of Bifidobacteria in Children Affected by Seasonal Allergic Rhinitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Michele Miraglia del Giudice, Prof. Associato, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRB01
Record Dates: First submitted 2016-06-10; First posted 2016-06-21 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifidobacteria mixture 0.5 ml (Active Comparator): Bifidobacteria 0.5 ml per os all days for 2 months
  Interventions: Drug: Bifidobacteria
- placebo (Placebo Comparator): Placebo 0.5 ml per os all days for 2 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bifidobacteria — 0.5 ml per os all days for 2 months
  Other Names: longum infantis M16V
  Arms: Bifidobacteria mixture 0.5 ml
Drug: placebo — 0,5 ml per os all days for 2 months
  Arms: placebo

SUMMARY:
This study is aimed at assessing the efficacy of supplementation with a mixture of three bifidobacteria , on the allergic rhinitis..The rhinitis symptoms were assessed by validated score ( TSS ) , for children aged between 4 and 17 years with allergic rhinitis parietaria , mild , moderate or severe , than children not supplemented .

Secondary Objectives

* The effectiveness of treatment by VAS :
* Evaluation of the rescue medication consumption
* Evaluation of quality of life ( using structured questionnaire )
* Evaluation of the frequency and school performance ( using structured questionnaire )
* Assessment of sleep quality and attention (through structured questionnaire )
* Satisfaction rating and satisfaction of parents
* Evaluation of asthma exacerbations in children susceptible

DETAILED DESCRIPTION:
This is a randomized , double-blind , placebo - controlled , phase 3 , 2 arms , in which patients were selected to receive placebo or a mixture powder composed of three bifidobacteria : Bifidobacterium Longum BB536 ( 3 billion units ) + Bifidobacterium infantis M - 63 ( 1 billion units ) Bifidobacterium breve M + -16 V ( 1 billion units ) . The subjects included in our study are represented by children aged between 4 and 17 years , with seasonal allergic rhinitis moderate and presenting positive skin prick test against parietaria.The participation of each subject in the study was based on evaluation of its clinical history. The recruited patients were divided into two groups according to the drug used.The group A received placebo , while the group B mixture bifidobacteria. The treatment was performed for a period of two months. At the beginning and at the end of therapy several surveys have been carried out , so as to be able to compare results and to draw some preliminary conclusions about the effectiveness of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes , aged from 4 to 17 years
* History seasonal allergic rhinitis mild , moderate or severe , according to the guidelines defined AIR 2013 , documented by recurrent episodes in the previous year and confirmed by skin prick test positive
* Written informed consent of one parent or a legal representative

Exclusion Criteria:

* Lack of written informed consent by at least one parent or a legal representative
* Concurrent disorders such as infection of the upper or lower respiratory tract , nasal surgery in the past year , respiratory tract abnormalities , immune diseases
* Use of antihistamines , nasal or systemic corticosteroids , leukotriene modifiers , or cromolyn sodium , on an ongoing basis used in the last six weeks.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the symptoms by structural questionary | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Second University, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miraglia Del Giudice M, Indolfi C, Capasso M, Maiello N, Decimo F, Ciprandi G. Bifidobacterium mixture (B longum BB536, B infantis M-63, B breve M-16V) treatment in children with seasonal allergic rhinitis and intermittent asthma. Ital J Pediatr. 2017 Mar 7;43(1):25. doi: 10.1186/s13052-017-0340-5. PMID 28270216